CLINICAL TRIAL: NCT01783028
Title: Home-Based Asthma Support and Education for Adults
Acronym: HomeBase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health - Seattle and King County (Other Government)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, James Krieger, Chief of Chronic Disease and Injury Prevention, Public Health - Seattle and King County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHSKC-AST-HomeBASE; 1R01ES014583-01A1 (NIH)
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Health Worker support (Experimental): home visits from community health workers providing education and support for self-management of asthma, assessment of the home for environmental triggers, resources for asthma control, and assistance in effective communication with medical providers
  Interventions: Behavioral: Community Health Worker support
- the usual care control group (No Intervention): Usual care is defined as services received by participants in the absence of the intervention plus information about community resources that support asthma self-management (such as classes and support groups) and educational pamphlets

INTERVENTIONS:
Behavioral: Community Health Worker support — For the intervention group, a trained Community Health Worker (CHW) provided education, support and service coordination through home visits. The CHW first made an in home assessment visit. At the assessment visit, the participant had the opportunity to ask questions and sign written consent. During this visit, the CHW assessed the participant's knowledge of asthma, current status of asthma control, challenges with controlling asthma, self-management practices and exposure to asthma triggers. After enrollment, the participant received up to four follow-up educational visits 0.5, 1.5, 3.5 and 7 months later. In addition to scheduled visits, the CHWs worked with their participants on an as-needed basis via telephone, email, or additional home visits.
  Other Names: CHW intervention
  Arms: Community Health Worker support

SUMMARY:
This study tests the hypothesis that community health workers providing home visits to provide education and support for self-management of asthma, assessment of the home for environmental triggers, resources for asthma control, and assistance in effective communication with medical providers over the course of one year would reduce asthma morbidity, asthma-related urgent health care use and exposure to indoor asthma triggers among low income adults with not well controlled asthma.

DETAILED DESCRIPTION:
We used a randomized controlled parallel group design to compare the intervention to a usual-care control group. We attempted to evaluate the effectiveness of the intervention in the "real world," rather than its ideal efficacy.

The CHWs used protocols that specified education content, participant skill development and participant and CHW actions. The CHWs modified their approach to meet the priorities of participants using motivational interviewing techniques. They addressed asthma patho-physiology, reliever and controller medication use, self-monitoring, use of an asthma action plan, environmental assessment, trigger avoidance, effective use of the health care system, successful communication with health care providers, and weight control (obesity is associated with increased asthma symptoms). Participants also received low-literacy educational materials, in English or Spanish. The education concepts and environmental assessment activities were based on our prior healthy homes work modified for adults.

ELIGIBILITY:
Inclusion Criteria:

* residence of King County Washington
* household income below the 250% of the 2007 federal poverty level
* had "not well controlled asthma" or "very poorly controlled asthma"

Exclusion Criteria:

* speak a language other than English or Spanish
* no permanent housing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2008-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
asthma symptom-free days during the last two weeks | baseline and 12 months after enrollment
  Asthma symptoms are evaluated using the following questions:
  1. During the past 14 days (that is, during the past fourteen 24 hour periods that include daytime and nighttime), on how many DAYS did you have any asthma symptoms, such as wheezing, coughing, tightness in the chest, shortness of breath, waking up at night because of asthma symptoms, or slowing down of usual activities because of asthma?
  2. During the DAYTIME in the past 14 days, how many DAYS did you have asthma symptoms, such as wheezing, cough, tightness in the chest, or shortness of breath?
  3. During the past 14 days, how many days did you have to slow down or stop your usual activities because of asthma, wheezing or tightness in the chest, or cough?
  4. During the NIGHTTIME in the past 14 nights, how many NIGHTS did you WAKE UP because of asthma, wheezing, cough, tightness in the chest, or shortness of breath?.

SECONDARY OUTCOMES:
Asthma-related quality of life score during the last two weeks | baseline and 12 months after enrollment
  Asthma Quality of Life Questionnaire
  http://www.qoltech.co.uk/aqlq.html

OTHER OUTCOMES:
health care utilization | baseline and 12 months after enrollment
  health care utilization includes asthma-related hospitalization, emergency department visit, and unscheduled clinic visit during the past 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James Krieger, MD, Principal Investigator — Public Health - Seattle and King County
Locations (1):
- Public Health - Seattle & King County, Seattle, Washington, United States

REFERENCES:
- [Derived] Krieger J, Song L, Philby M. Community health worker home visits for adults with uncontrolled asthma: the HomeBASE Trial randomized clinical trial. JAMA Intern Med. 2015 Jan;175(1):109-17. doi: 10.1001/jamainternmed.2014.6353. PMID 25419871